CLINICAL TRIAL: NCT03600298
Title: Does Simulation Enhance Closed-Loop Communication in the Clinical Setting of a Pediatric Intensive Care Unit?
Brief Title: Simulation Training of Closed-Loop Communication (CLC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ulmer-Riva2017
Record Dates: First submitted 2018-06-28; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Pediatric Intensive Care Unit; Closed Loop Communication; In-situ Simulation; Behavioral Changes
MeSH Terms: conditions — Teach-Back Communication

STUDY DESIGN:
Intervention Model Description: Open interventional before and after study on the effect of on-site full-scale simulation with a subsequent course follow-up and a three month follow-up observation pertaining to behavioural changes in communication of the paediatric intensive care unit staff that is participating in the on-site simulation training
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric intensive care unit-nurses (Other): Phase I: During the month leading up to the simulation two trained observers / raters will observe the rate of Closed-Loop Communication in the pediatric intensive care unit (PICU) among study participants.
  Intervention phase: Study participants will be subjected to on-site simulation training focusing on communication, including CRM and non-technical skills in the PICU setting.
  Phase II + III: During the follow up phase, trained raters will again observe the study-participating PICU staff relative to their communication behaviour in the month following simulation training (Phase II) and again three months later (Phase III).
  Interventions: Other: Simulation

INTERVENTIONS:
Other: Simulation — Intervention phase: Study participants will be subjected to on-site simulation training focusing on communication, including CRM and non-technical skills in the PICU setting.

SUMMARY:
Open interventional before and after study on the effect of on-site full-scale simulation with a subsequent course follow-up and a three month follow-up observation pertaining to behavioural changes in communication of the paediatric intensive care unit staff that is participating in the on-site simulation training.

DETAILED DESCRIPTION:
Closed-Loop Communication (CLC) is a proposed, taught and practiced Crisis Resource Management (CRM) strategy thought to be effective for enhancing patient safety by enforcing reiteration and clarity, thus reducing ambiguity during verbal communication among health care providers. The transfer of this CRM strategy into clinical practice seems to require recurring exposure. Teaching and training is needed to help health care providers develop routine in communicating. This training is most effective if practiced in the clinical setting that is familiar to the health care provider (in situ simulation). As trainees become more proficient, the ultimate goal is to integrate Closed-Loop Communication into daily habits of verbal interaction in every health care setting. One way to practice the utilization of Closed-Loop Communication is simulation. The investigators seek to investigate if simulation participants can incorporate CRM strategies such as Closed-Loop Communication into their communication repertoire. This shall serve as an example of attitude transfer following a simulation based learning experience.The primary study objective is to measure the success of simulation training for increasing Closed-Loop Communication as a behavioural change in the clinical setting.

ELIGIBILITY:
Inclusion criteria:

* Employees, with written informed consent, working in the paediatric intensive care unit of the Children's Bern University Hospital
* Employees novices to in-situ simulation

Exclusion criteria:

* employees, working in the paediatric intensive care unit of the Children's Bern University Hospital who are not fluent in German or Swiss German.
* employees, working in the paediatric intensive care unit of the Children's Bern University Hospital who are unable to be observed during phases I and II and during the follow up phase (see below).
* No vulnerable participants will be included.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
Measurement of difference regarding employment of Closed-Loop communications measured by counting the call-outs for each participant in a defined timeframe in Phase I, II and III of the study | 3 months
  measurement of difference regarding the employment of Closed-Loop Communication in the clinical setting after three months of the simulation training focusing on crisis resource management (CRM) in communication and assessed by external raters and compared to baseline before such training. Based on a study by Härgestam et al. (2013) we classified the call-outs as command (com), question (que), observation (obs) or suggestion (sug). Furthermore, after our experience during the pilot phase we added the category information (inf), since we could not sort a number of call-outs into the existing four categories

SECONDARY OUTCOMES:
Rate of Closed-Loop Communication measured by counting the call-outs for each participant in a defined timeframe in Phase I, II and III of the study | 3 months
  rate of Closed-Loop Communication following the simulation as assessed by external raters
Measurement of difference regarding employment of Closed-Loop communications measured by counting the reaction to call-outs for each participant in a defined timeframe in Phase I, II and III of the study | 3 months
  measurement of difference regarding the employment of Closed-Loop Communication while reacting to a call-outs in the clinical setting after three months of the simulation training focusing on crisis resource management (CRM) in communication and assessed by external raters and compared to baseline before such training. Inspired by the study by Boyd et al (2014) the reaction to the call-out will be as follows categorized: no response (no-check), call-back (check), verbal response (verb-res.), nonverbal response (noverb-res.) and closed-loop (check-close).
Rate of Closed-Loop Communication measured by counting the reactions to call-outs for each participant in a defined timeframe in Phase I, II and III of the study | 3 months
  rate of Closed-Loop Communication following the simulation as assessed by external raters

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Riva, MD, Study Director — University of Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Derived] Ulmer FF, Lutz AM, Muller F, Riva T, Butikofer L, Greif R. Communication Patterns During Routine Patient Care in a Pediatric Intensive Care Unit: The Behavioral Impact of In Situ Simulation. J Patient Saf. 2022 Mar 1;18(2):e573-e579. doi: 10.1097/PTS.0000000000000872. PMID 34224500